CLINICAL TRIAL: NCT06554405
Title: Examining the Effects of Bilateral Neuromobilization in Patients With Carpal Tunnel Syndrome: Comparison Study With Unilateral Application
Brief Title: Bilateral vs. Unilateral Neuromobilization in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Öznur Güney, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GaziU-GUNEY-001
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Neuromobilization; Median Nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be grouped according to randomization into unilateral or bilateral intervention.
Who Masked: Outcomes Assessor
Masking Description: The researcher who will evaluate the patients before and after treatment will not know which group the patients are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Intervention (Active Comparator): Patients will be treated for 4 weeks (2 days in a week, 8 sessions). The treatment plan involves massage therapy, neuromobilization exercises and cold application. In this arm, treatment plan will be applied only for the symptomatic side. The rest of the treatment will be the same as the other group.
  Interventions: Other: Unilateral Intervention
- Bilateral Intervention (Experimental): Patients will be treated for 4 weeks (2 days in a week, 8 sessions). The treatment plan involves massage therapy, neuromobilization exercises and cold application. In this arm, treatment plan will be applied only for both symptomatic and nonsymptomatic sides. The rest of the treatment will be the same as the other group.
  Interventions: Other: Bilateral Intervention

INTERVENTIONS:
Other: Unilateral Intervention — Treatment plan will be applied to the symptomatic side.
  Arms: Unilateral Intervention
Other: Bilateral Intervention — Treatment plan will be applied to the symptomatic and nonsymptomatic sides.
  Arms: Bilateral Intervention

SUMMARY:
This study aims to investigate whether bilateral (both extremities together) neuromobilization is superior to unilateral (only the affected side) neuromobilization in individuals diagnosed with Carpal Tunnel Syndrome.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome (CTS) is defined as an upper extremity nerve entrapment resulting from the compression of the median nerve at the wrist level. It is the most common entrapment neuropathy. Patients with CTS experience numbness, tingling, and pain in the hand, which can sometimes extend to the arm, along with hand weakness and thenar atrophy. These symptoms typically worsen after hand use and at night. While clinical findings are absent in the early stages of the disease, sensory and strength loss is observed in the areas innervated by the median nerve in advanced stages.

The pathophysiology of CTS includes hypertrophic changes in the synovial tissue of the flexor tendon, connective tissue changes in the median nerve, conduction disturbances, and increased pressure in the carpal tunnel.

Treatment is tailored to the patient's symptoms. Conservative treatment is preferred in mild to moderate stages, while surgical intervention may be necessary in advanced stages. All patients should receive education on ergonomics aimed at reducing symptoms in daily life.

Conservative treatment for CTS includes nerve mobilization techniques, the use of orthoses to maintain the wrist in a neutral position, electrotherapy (ESWT, laser), manual therapy, kinesiotaping, corticosteroid and platelet-rich plasma (PRP) injections, and anti-inflammatory medications. Patients who do not respond to conservative treatment are referred for surgery.

Neural structures are capable of tolerating significant tension and compression forces encountered during daily activities and sports. This capability is due to the connective tissue sheath surrounding the nerve.

The musculoskeletal system creates an environment that surrounds the nervous system, and its movements affect peripheral nerves. With the excursion (sliding) movement, compression on the peripheral nerve decreases. Clinical neuromobilization is a manual therapy method that integrates the mechanics and physiology of the nervous system with musculoskeletal function. Neuromobilization (NM) aims to balance the relationship between neural tissues and surrounding mechanical tissues, thereby regulating optimal physiological functions.

The aim of using neuromobilization exercises with sliding techniques in nerve entrapments is to increase axonal transport and improve nerve conduction. It has been suggested that these exercises can reduce pressure within the nerve, improve its blood supply, and thus contribute to nerve regeneration. Recent studies in the literature report that neuromobilization exercises have supportive effects in pain improvement, reduction of distal latency time, and increased pinch strength. A systematic review indicated these effects as pain improvement, lowering the pain threshold, improving function, and avoiding surgery. It was stated that neuromobilization exercises added to the CTS treatment program accelerate the rehabilitation process and enhance recovery.

Although there are studies in the literature proving the superiority of neuromobilization over other treatment methods, the number of studies investigating the application of neuromobilization to the unaffected side is limited. Considering that the connective tissue sheaths surrounding peripheral nerves in both upper extremities are connected via the central nervous system, it is hypothesized that neuromobilization applied to the unaffected side or bilaterally might be more effective on the symptomatic side compared to unilateral application. However, studies that consider this connection and include the unaffected side in treatment are significantly lacking.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with CTS,
* Aged 18 and above,
* Without any other conditions in either upper extremity (such as trigger finger, osteoarthritis, tenosynovitis)

Exclusion Criteria:

* Individuals with a history of surgery, trauma, or fracture in the same upper extremity,
* Those who have received an injection for CTS in the last 3 months,
* Those with poor cooperation,
* Those participating in any other treatment program during the study,
* Those with a history of uncontrolled systemic diseases or systemic diseases involved in the etiology of CTS (such as diabetes, thyroid diseases, rheumatoid arthritis),
* Those who have used orthoses regularly and/or received physiotherapy in the last 3 months,
* Individuals with marked thenar atrophy requiring early surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Symptom Severity Assessment (Boston Carpal Tunnel Syndrome Questionnaire- Symptom Severity Scale) | Four weeks
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ), developed in 1993, will be used to assess individuals' functional status and symptoms. The Turkish validity and reliability study of the test has been conducted. The test consists of two self-assessment sections: one with 11 questions evaluating symptom severity and another with 8 questions evaluating functional capacity. It is a Likert-type questionnaire, where 1 indicates the best condition and 5 indicates the worst condition. The total score is calculated by dividing the total points by the number of questions, resulting in a score between 1 and 5.

SECONDARY OUTCOMES:
Light Touch and Pressure Sense | Four weeks
  Light touch and pressure assessment will be performed using the Semmes-Weinstein Monofilament test. This test kit contains five filaments ranging from 2.83 (0.07 grams of force) to 6.65 (300 grams of force). These filaments are applied to the skin. During the assessment, the individual should not see the filament. First, the unaffected side is assessed, followed by the affected side. During the evaluation, the filament is applied to the skin at a 90-degree angle and held for 1.5 seconds. The application sites for the median nerve are the pulp of the first finger and the pulp of the second finger. The patient is asked if they can feel the filament and should respond with "yes" or "no." The evaluation starts with the lowest filament, 2.83, which represents normal sensation. If the patient responds "yes," their sensation is recorded as normal. If not, progressively higher-value filaments are used until a "yes" response is obtained.
Visual Analog Scale (VAS) | Four weeks
  The Visual Analog Scale (VAS) will be used for pain assessment. The individual will make a mark on a 10-centimeter horizontal line, where 0 indicates no pain and 10 indicates maximum pain. This marking will be done separately for both rest and activity periods. The data will be recorded in centimeters.
Gross Grip Strength | Four weeks
  For gross grip strength measurement, a hydraulic hand dynamometer (Baseline®, USA) will be used. The measurement will be conducted in the standard position specified by the American Society of Hand Therapists. In this position, the individual will sit on a chair with back support, with the elbow at 90 degrees of flexion and the wrist in a neutral position. The person will be asked to squeeze the dynamometer with maximum force. The measurement will be repeated three times, and the average will be recorded in kg/f.
Pinch Grip Strength | Four weeks
  For pinch grip strength measurement, a mechanical pinch meter (Baseline®, USA) will be used. Lateral (key) pinch, two-point (bipod, tip) pinch, and three-point (tripod, palmar) pinch measurements will be performed separately. For the lateral pinch, the patient will be asked to squeeze the end of the pinch meter between the thumb and the lateral surface of the middle phalanx of the second finger with maximum force. For the two-point pinch strength measurement, the patient will be asked to squeeze the pinch meter between the thumb and the pulp of the second finger, and for the three-point pinch strength measurement, between the thumb, the second finger, and the third finger as tightly as possible. Assessments will be conducted bilaterally, starting with the healthy side. The measurements will be repeated three times for each side, and the averages will be recorded in kg/f.
Functional Level Assessment (Boston Carpal Tunnel Syndrome Questionnaire-Functional Status Scale) | Four weeks
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ), developed in 1993, will be used to assess individuals' functional status and symptoms. The Turkish validity and reliability study of the test has been conducted. The test consists of two self-assessment sections: one with 11 questions evaluating symptom severity and another with 8 questions evaluating functional capacity. It is a Likert-type questionnaire, where 1 indicates the best condition and 5 indicates the worst condition. The total score is calculated by dividing the total points by the number of questions, resulting in a score between 1 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Öznur GÜNEY, Study Chair — Zonguldak Bulent Ecevit University
Locations (1):
- Gazi University Faculty of Health Sciences, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No